CLINICAL TRIAL: NCT03818256
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Efficacy, and Pharmacokinetics of Miricorilant (CORT118335) in Obese Adult Patients With Schizophrenia or Bipolar Disorder and Recent Weight Gain While Taking Antipsychotic Medications (GRATITUDE)
Brief Title: A Study to Assess the Safety, Efficacy, and Pharmacokinetics of Miricorilant (CORT118335) in Obese Adults With Schizophrenia or Bipolar Disorder Treated With Antipsychotic Medications
Acronym: GRATITUDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CORT118335-876
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Antipsychotic-induced Weight Gain (AIWG)
Keywords: Antipsychotic-induced weight gain (AIWG); Obesity; Weight Gain; Mental disorders; Schizophrenia; Risperidone; Quetiapine; Olanzapine; Bipolar Disorder
MeSH Terms: conditions — Obesity; Weight Gain; Mental Disorders; Schizophrenia; Bipolar Disorder | interventions — CORT118335

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Miricorilant 600 mg (Experimental): Patients who meet the entry criteria will be randomized to receive 600 mg miricorilant for 12 weeks.
  Interventions: Drug: Miricorilant
- Placebo (Placebo Comparator): Patients who meet the entry criteria will be randomized to receive placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Miricorilant — Miricorilant 600 mg (6 X 100 mg tablets) for once-daily oral dosing
  Other Names: CORT118335
  Arms: Miricorilant 600 mg
Drug: Placebo — Placebo tablets for once-daily oral dosing
  Arms: Placebo

SUMMARY:
This phase 2, double blind, placebo-controlled, randomized study is to assess the safety, efficacy, and pharmacokinetics (PK) of miricorilant (CORT118335) in obese adults with schizophrenia or bipolar disorder treated with antipsychotic medications.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study that will assess the safety, efficacy, and PK of miricorilant in obese patients with schizophrenia or bipolar disorder who are currently taking oral or injectable atypical antipsychotic medication.

Patients who meet the criteria for the Study CORT118335-876 will be randomized on Day 1 to receive 600 mg miricorilant or placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of schizophrenia or bipolar disorder
* Are currently taking oral or injectable atypical antipsychotic medication (except clozapine) and must have documented weight gain while on these medications
* Must be on a stable dose of medication for 1 month prior to Screening
* Are able to successfully complete placebo tablet swallow test
* Have a BMI ≥30 kg/m^2.

Exclusion Criteria:

* Have a history of a medical condition affecting body weight (eg, poorly controlled hyper- or hypothyroidism; eating disorder such as anorexia, bulimia, or binge eating; or polycystic ovary syndrome)
* Have poorly controlled diabetes mellitus
* Have poorly controlled hypertension
* Have a history of symptomatic hypotension
* Have a history of orthostatic hypotension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Juneja, MD, Study Director — Corcept Therapeutics
Locations (26):
- United States (26):
  - Site 143, Bentonville, Arkansas
  - Site 249, Little Rock, Arkansas
  - Site 153, Culver City, California
  - Site 239, Garden Grove, California
  - Site 134, Lemon Grove, California
  - Site 126, Oakland, California
  - Site 163, Oceanside, California
  - Site 229, Rancho Cucamonga, California
  - Site 202, Miami, Florida
  - Site 144, North Miami, Florida
  - Site 241, Okeechobee, Florida
  - Site 140, Chicago, Illinois
  - Site 140, Lincolnwood, Illinois
  - Site 146, Wichita, Kansas
  - Site 138, Glen Burnie, Maryland
  - Site 151, Las Vegas, Nevada
  - Site 216, New York, New York
  - Site 181, Raleigh, North Carolina
  - Site 107, Dayton, Ohio
  - Site 235, Thorndale, Pennsylvania
  - Site 235, West Chester, Pennsylvania
  - Site 206, DeSoto, Texas
  - Site 066, Houston, Texas
  - Site 165, Richardson, Texas
  - Site 139, Salt Lake City, Utah
  - Site 137, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients who meet the entry criteria will be randomized to receive placebo for 12 weeks.
  Placebo: Placebo tablets for once daily oral dosing
Period: Overall Study
Arm/Group | Miricorilant 600 mg | Placebo
Started | 35 | 36
Completed | 27 | 28
Not Completed | 8 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 0 | 5
Not completed — Gaining weight without prohibited medication vyvanse | 1 | 0
Not completed — Not reporting for scheduled visits | 1 | 0
Not completed — Non-compliant with investigational product | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Miricorilant 600 mg | Placebo | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (10.50) | 47.5 (11.78) | 45.7 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 16 | 29
  White | 21 | 20 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 36 | 71
Body weight [Mean (Standard Deviation); unit: kg] | 110.39 (20.01) | 107.69 (25.41) | 109.02 (22.79)
Homeostatic model assessment for insulin resistance (HOMA-IR) [Mean (Standard Deviation); unit: HOMA-IR score] — HOMA-IR = [fasting plasma glucose (mg/dL) X fasting insulin (µU/mL)]/405. HOMA-IR is a method to evaluate insulin sensitivity. The HOMA-IR score should be ≤1.0 to be considered normal. A score >1.9 indicates early insulin resistance and a score >2.9 indicates significant insulin resistance. Population: Two patients in the placebo group did not have a Baseline HOMA-IR measurement.
  HOMA-IR score
    number analyzed (Participants) | 35 | 34 | 69
    (all) | 8.687 (5.71) | 8.463 (17.27) | 8.577 (13.24)
Waist-to-hip ratio [Mean (Standard Deviation); unit: Ratio] — Waist-to-hip ratio compares the circumference of the waist to the circumference of the hips. The ratio is calculated by dividing the waist measurement by the hip measurement, using the same units of measurement for both. A waist-to-hip ratio <0.95 in men and <0.80 in women is considered healthy.
  Ratio | 1.032 (0.24) | 0.967 (0.10) | 0.999 (0.18)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Weight at Week 12 for 600 mg Miricorilant Versus Placebo
Time Frame: Baseline Day 1 and Week 12
Population: The Efficacy Evaluable Population was patients who received ≥4 weeks of study drug and had body weight assessed at Baseline and on Week 12.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Miricorilant 600 mg | Placebo
Number analyzed (Participants) | 29 | 29
kg | -0.98 (0.414) | -1.08 (0.415)
Statistical Analysis 1: Comparison: Miricorilant 600 mg vs Placebo; Test type: Superiority; p = 0.8511, Mixed Models Analysis; Least Squares Mean Difference = 0.11, 95% CI 2-sided [-1.03 to 1.24]

2. Primary Outcome: Number of Patients With One or More Treatment-emergent Adverse Events
Time Frame: Up to Follow-up Visit (Week 16)
Population: The Safety Population included patients who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Miricorilant 600 mg | Placebo
Number analyzed (Participants) | 35 | 36
Participants | 16 | 18

3. Primary Outcome: Number of Patients With One or More Treatment-emergent Serious Adverse Events
Time Frame: Up to Follow-up Visit (up to Week 16)
Population: The Safety Population included patients who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Miricorilant 600 mg | Placebo
Number analyzed (Participants) | 35 | 36
Participants | 1 | 1

4. Primary Outcome: Number of Patients With One or More Treatment-emergent Adverse Events Leading to Early Study Discontinuation
Time Frame: Up to Follow-up Visit (up to Week 16)
Population: The Safety Population included patients who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Miricorilant 600 mg | Placebo
Number analyzed (Participants) | 35 | 36
Participants | 3 | 1

5. Secondary Outcome: Percentage of Patients Achieving More Than or Equal to 5% Weight Loss
Time Frame: Baseline Day 1 to Week 12
Population: The Efficacy Evaluable Population was patients who received ≥4 weeks of study drug and had baseline and ≥1 body weight measurement taken on or after Week 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Miricorilant 600 mg | Placebo
Number analyzed (Participants) | 33 | 33
Participants | 2 | 3
Statistical Analysis 1: Comparison: Miricorilant 600 mg vs Placebo; Test type: Superiority; p = 0.8169, Regression, Logistic; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.150 to 4.474]

6. Secondary Outcome: Change From Baseline in HOMA-IR at Week 12
Description: HOMA-IR = [fasting plasma glucose (mg/dL) X fasting insulin (µU/mL)]/405. HOMA-IR is a method to evaluate insulin sensitivity. The HOMA-IR score should be ≤1.0 to be considered normal. A score >1.9 indicates early insulin resistance and a score >2.9 indicates significant insulin resistance.
Time Frame: Baseline Day 1 and Week 12
Population: The Efficacy Evaluable Population was patients who received ≥4 weeks of study drug and had HOMA-IR assessed at Baseline and on Week 12.
Measure: Median (Inter-Quartile Range); unit: HOMA-IR score
Arm/Group | Miricorilant 600 mg | Placebo
Number analyzed (Participants) | 26 | 23
HOMA-IR score | 1.080 [-2.020 to 3.780] | 0.890 [-0.970 to 2.400]
Statistical Analysis 1: Comparison: Miricorilant 600 mg vs Placebo; Test type: Superiority; p = 0.9285, Wilcoxon rank-sum test; Location shift = 0.175, 95% CI 2-sided [-2.860 to 2.780]

7. Secondary Outcome: Change From Baseline in Waist-to-hip Ratio at Week 12
Description: Waist-to-hip ratio compares the circumference of the waist to the circumference of the hips. The ratio is calculated by dividing the waist measurement by the hip measurement, using the same units of measurement for both. A waist-to-hip ratio <0.95 in men and <0.80 in women is considered healthy.
Time Frame: Baseline Day 1 and Week 12
Population: The Efficacy Evaluable Population was patients who received ≥4 weeks of study drug and had hip and waist measurements at Baseline and on Week 12.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Miricorilant 600 mg | Placebo
Number analyzed (Participants) | 29 | 29
Ratio | 0.008 (0.0092) | 0.001 (0.0091)
Statistical Analysis 1: Comparison: Miricorilant 600 mg vs Placebo; Test type: Superiority; p = 0.5669, Mixed Models Analysis; Least squares mean difference = 0.007, 95% CI 2-sided [-0.018 to 0.033]

ADVERSE EVENTS:
Time Frame: Baseline Day 1 to Week 16
Description: The Safety Population included patients who received ≥1 dose of study drug.
Arm/Group | Miricorilant 600 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/35 | 1/36
Other Adverse Events (participants affected / at risk) | 12/35 | 5/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Miricorilant 600 mg (N=35) | Placebo (N=36)
Hyperthermia malignant (General disorders) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Mania (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Miricorilant 600 mg (N=35) | Placebo (N=36)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Alanine aminotransferase increased (Investigations) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 1
Akathisia (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual publications will be allowed before publication of the multicenter results except as agreed with Corcept. The Investigator agrees to submit all manuscripts or abstracts to Corcept for review before submission to the publisher.

DOCUMENTS (2):
  • Study Protocol (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT03818256/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT03818256/SAP_001.pdf